CLINICAL TRIAL: NCT04362085
Title: Coagulopathy of COVID-19: A Pragmatic Randomized Controlled Trial of Therapeutic Anticoagulation Versus Standard Care as a Rapid Response to the COVID-19 Pandemic (RAPID COVID COAG)
Brief Title: Coagulopathy of COVID-19: A Pragmatic Randomized Controlled Trial of Therapeutic Anticoagulation Versus Standard Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Vermont Medical Center (Other); University of Sao Paulo (Other); Hopital Charles Lemoyne (Other); William Osler Health System (Other); MOUNT SINAI HOSPITAL (Other); Trillium Health Partners (Other); St. Joseph's Health Centre Toronto (Other); The Ottawa Hospital (Other); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other); Michael Garron Hospital (Other); University of Alberta (Other); Southlake Regional Health Centre (Other); Maisonneuve-Rosemont Hospital (Other); Queen Elizabeth II Health Sciences Centre (Other); Foothills Medical Centre (Other); Alberta Health services (Other); Peter Lougheed Centre (Other); Mater Misericordiae University Hospital (Other); King Saud Medical City (Other Government); King Fahad Medical City (Other Government); King Faisal Specialist Hospital & Research Center (Other); Versiti Blood Health (Other); Barnes-Jewish Hospital (Other); Al Ain Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAPID COVID-COAG
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-08

CONDITIONS: COVID-19
Keywords: coagulopathy; anticoagulation
MeSH Terms: conditions — COVID-19; Hemostatic Disorders

STUDY DESIGN:
Intervention Model Description: This study is a 2-arm, parallel, pragmatic, multi-centre, open-label randomized controlled trial to determine the effect of therapeutic anticoagulation on the composite outcome of ICU admission, mechanical ventilation and/or death in hospitalized patients with COVID-19.
Masking Description: Blinding of participants, clinical research staff, and clinicians is not possible due to the nature of the intervention. However, the biostatisticians will be blinded at the data analysis phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Anticoagulation (Experimental): Therapeutic anticoagulation with LMWH or UFH (high dose nomogram). The choice of LMWH versus UFH will be at the clinician's discretion and dependent on local institutional supply. Therapeutic anticoagulation will be administered until discharged from hospital, 28 days or death. If the patient is admitted to the ICU or requiring ventilatory support, we recommend continuation of the allocated treatment as long as the treating physician is in agreement.
  Interventions: Drug: Therapeutic Anticoagulation
- Standard Care (No Intervention): Administration of LMWH, UFH or fondaparinux at thromboprophylactic doses for acutely ill hospitalized medical patients, in the absence of contraindication, is considered standard care.

INTERVENTIONS:
Drug: Therapeutic Anticoagulation — The choice of low molecular weight heparin (LMWH) versus unfractionated heparin (UFH) will be at the clinician's discretion. LMWH options include: Tinzaparin, Enoxaparin or Dalteparin. UFH will be administered using a weight-based nomogram with titration according to center-specific institutional protocol.
  Arms: Therapeutic Anticoagulation

SUMMARY:
Coagulopathy of COVID-19 afflicts approximately 20% of patients with severe COVID-19 and is associated with need for critical care and death. COVID-19 coagulopathy is characterized by elevated D-dimer, an indicator of fibrin formation and clot lysis, and a mildly prolonged prothrombin time, suggestive of coagulation consumption. To date, it seems that COVID-19 coagulopathy manifests with thromboembolism, thus anticoagulation may be of benefit. We propose to conduct a parallel pragmatic multi-centre open-label randomized controlled trial to determine the effect of therapeutic anticoagulation compared to standard care in hospitalized patients admitted for COVID-19 with an elevated D-dimer.

DETAILED DESCRIPTION:
2-arm, parallel, pragmatic, multi-centre, open-label randomized controlled trial to determine the effect of therapeutic anticoagulation, with low molecular weight heparin or unfractionated heparin (high dose nomogram), compared to standard care in hospitalized patients with COVID-19 and an elevated D-dimer on the composite outcome of intensive care unit (ICU) admission, non-invasive positive pressure ventilation, invasive mechanical ventilation or death at 28 days. Eligible participants will be randomized to one of two treatment regimens, receiving either therapeutic anticoagulation or standard care until discharged from hospital, death or day 28.

The primary composite outcome of ICU admission, non-invasive positive pressure ventilation, invasive mechanical ventilation, or all-cause death up to 28 days.

Key secondary outcomes between study arms up to day 28 include:

1. All-cause death
2. Composite outcome of ICU admission or all-cause death
3. Composite outcome of mechanical ventilation or all-cause death
4. Major bleeding as defined by the ISTH Scientific and Standardization Committee (ISTH-SSC) recommendation
5. Number of participants who received red blood cell transfusion (≥1 unit)
6. Number of participants with transfusion of platelets, frozen plasma, prothrombin complex concentrate, cryoprecipitate and/or fibrinogen concentrate
7. Renal replacement therapy;
8. Number of hospital-free days alive
9. Number of ICU-free days alive
10. Number of ventilator-free days alive
11. Number of organ support-free days alive
12. Number of participants with venous thromboembolism
13. Number of participants with arterial thromboembolism
14. Number of participants with heparin induced thrombocytopenia
15. Changes in D-dimer up to day 3

The treatment arm is therapeutic anticoagulation with low molecular weight heparin (LMWH) or unfractionated heparin (UFH, high dose nomogram). The choice of LMWH versus UFH will be at the clinician's discretion. LMWH options include: Tinzaparin, Enoxaparin, or Dalteparin. UFH will be administered using a weight-based nomogram with titration according to the center-specific protocol. Therapeutic anticoagulation will be administered until discharged from hospital, 28 days or death. If the patient is admitted to the ICU or requiring ventilatory support, we recommend continuation of the allocated treatment as long as the treating physician is in agreement. The standard care arm is the administration of LMWH, UFH or fondaparinux at thromboprophylactic doses in the absence of contraindication.

No study specific bloodwork will be ordered aside from a single D-dimer test (if not collected through standard of care) up to and including day 3 after randomization for all participants in both study arms. In those on the active treatment arm who are receiving UFH, the aPTT or UFH anti-Xa will be drawn according to local institutional UFH nomogram protocol guidance. All laboratory results will be collected from standard of care from admission to hospital discharge, death or 28 days, where available. An optional biobanking component will collect blood at baseline and 2 follow up time points.

This study will immediately impact the clinical care of patients with severe COVID-19 internationally, whether the findings are positive or negative, as COVID-19 coagulopathy is a highly prevalent complication of severe COVID-19 and may precede the respiratory manifestations that characterize it.

ELIGIBILITY:
The inclusion criteria are:

1. laboratory confirmed diagnosis of SARS-CoV-2 via reverse transcriptase polymerase chain reaction as per the World Health Organization protocol or by nucleic acid based isothermal amplification.Positive test prior to hospital admission OR within first 5 days (i.e. 120 hours) after hospital admission;
2. admitted to hospital for COVID-19;
3. one D-dimer value above ULN (5 days (i.e. 120 hours) of hospital admission) and either: a) D-Dimer ≥2 times ULN; or b) D-dimer above ULN and oxygen saturation ≤ 93% on room air;
4. ≥18 years of age;
5. informed consent from the patient (or legally authorized substitute decision maker).

The exclusion criteria are:

1. pregnancy;
2. hemoglobin <80 g/L in the last 72 hours;
3. platelet count <50 x 10^9/L in the last 72 hours;
4. known fibrinogen <1.5 g/L (if testing deemed clinically indicated by the treating physician prior to the initiation of anticoagulation);
5. known INR >1.8 (if testing deemed clinically indicated by the treating physician prior to the initiation of anticoagulation);
6. patient already on intermediate dosing of LMWH that cannot be changed (determination of what constitutes an intermediate dose is to be at the discretion of the treating clinician taking the local institutional thromboprophylaxis protocol for high risk patients into consideration);
7. patient already on therapeutic anticoagulation at the time of screening (low or high dose nomogram UFH, LMWH, warfarin, direct oral anticoagulant (any dose of dabigatran, apixaban, rivaroxaban, edoxaban);
8. patient on dual antiplatelet therapy, when one of the agents cannot be stopped safely;
9. known bleeding within the last 30 days requiring emergency room presentation or hospitalization;
10. known history of a bleeding disorder of an inherited or active acquired bleeding disorder;
11. known history of heparin-induced thrombocytopenia;
12. known allergy to UFH or LMWH;
13. admitted to the intensive care unit at the time of screening;
14. treated with non-invasive positive pressure ventilation or invasive mechanical ventilation at the time of screening (of note: high flow oxygen delivery via nasal cannula is acceptable and is not an exclusion criterion).
15. imminent death according to the judgement of the most responsible physician
16. enrollment in another clinical trial of antithrombotic therapy involving pre-intensive care unit hospitalized patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Sholzberg, MD, FRCPC, Principal Investigator — Unity Health Toronto; Peter Jüni, MD, FESC, Principal Investigator — Unity Health Toronto; Mary Cushman, MD, Principal Investigator — University of Vermont Medical Center, Vermont
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Sholzberg M, Tang GH, Rahhal H, AlHamzah M, Kreuziger LB, Ainle FN, Alomran F, Alayed K, Alsheef M, AlSumait F, Pompilio CE, Sperlich C, Tangri S, Tang T, Jaksa P, Suryanarayan D, Almarshoodi M, Castellucci LA, James PD, Lillicrap D, Carrier M, Beckett A, Colovos C, Jayakar J, Arsenault MP, Wu C, Doyon K, Andreou ER, Dounaevskaia V, Tseng EK, Lim G, Fralick M, Middeldorp S, Lee AYY, Zuo F, da Costa BR, Thorpe KE, Negri EM, Cushman M, Juni P; RAPID trial investigators. Effectiveness of therapeutic heparin versus prophylactic heparin on death, mechanical ventilation, or intensive care unit admission in moderately ill patients with covid-19 admitted to hospital: RAPID randomised clinical trial. BMJ. 2021 Oct 14;375:n2400. doi: 10.1136/bmj.n2400. PMID 34649864
- [Derived] Sholzberg M, Tang GH, Rahhal H, AlHamzah M, Kreuziger LB, Ni Ainle F, Alomran F, Alayed K, Alsheef M, AlSumait F, Pompilio CE, Sperlich C, Tangri S, Tang T, Jaksa P, Suryanarayan D, Almarshoodi M, Castellucci L, James PD, Lillicrap D, Carrier M, Beckett A, Colovos C, Jayakar J, Arsenault MP, Wu C, Doyon K, Andreou ER, Dounaevskaia V, Tseng EK, Lim G, Fralick M, Middeldorp S, Lee AYY, Zuo F, da Costa BR, Thorpe KE, Negri EM, Cushman M, Juni P; RAPID Trial investigators. Heparin for Moderately Ill Patients with Covid-19. medRxiv [Preprint]. 2021 Jul 12:2021.07.08.21259351. doi: 10.1101/2021.07.08.21259351. PMID 34268513
- [Derived] Sholzberg M, Tang GH, Negri E, Rahhal H, Kreuziger LB, Pompilio CE, James P, Fralick M, AlHamzah M, Alomran F, Tseng E, Lim G, Lillicrap D, Carrier M, Ainle FN, Beckett A, da Costa BR, Thorpe K, Middeldorp S, Lee A, Cushman M, Juni P. Coagulopathy of hospitalised COVID-19: A Pragmatic Randomised Controlled Trial of Therapeutic Anticoagulation versus Standard Care as a Rapid Response to the COVID-19 Pandemic (RAPID COVID COAG - RAPID Trial): A structured summary of a study protocol for a randomised controlled trial. Trials. 2021 Mar 10;22(1):202. doi: 10.1186/s13063-021-05076-0. PMID 33691765
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Therapeutic Anticoagulation | Standard Care
Started | 228 | 237
Completed | 228 | 237
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapeutic Anticoagulation | Standard Care | Total
Number analyzed (Participants) | 228 | 237 | 465
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (14.1) | 59.6 (15.5) | 60.0 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 96 | 201
  Male | 123 | 141 | 264
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  European | 97 | 96 | 193
  Middle Eastern, North African | 65 | 67 | 132
  Asian | 27 | 38 | 65
  Black or African American | 18 | 23 | 41
  Hispanic or Latino | 14 | 10 | 24
  American Indian, Alaska Native, First Nations, Indigenous/Aboriginal, Metis | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Missing Data | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Composite Outcome of ICU Admission, Non-invasive Positive Pressure Ventilation, Invasive Mechanical Ventilation, or All-cause Death up to 28 Days.
Description: Composite outcome of ICU admission, non-invasive positive pressure ventilation, invasive mechanical ventilation, or all-cause death up to 28 days.
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Anticoagulation | Standard Care
Number analyzed (Participants) | 228 | 237
Participants | 37 | 52

2. Secondary Outcome: All-cause Death
Description: All-cause death
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Anticoagulation | Standard Care
Number analyzed (Participants) | 228 | 237
Participants | 4 | 18

3. Secondary Outcome: Composite Outcome of ICU Admission or All-cause Death
Description: Composite outcome of ICU admission or all-cause death
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Anticoagulation | Standard Care
Number analyzed (Participants) | 228 | 237
Participants | 4 | 1

4. Secondary Outcome: Composite Outcome of Mechanical Ventilation or All-cause Death
Description: Composite outcome of mechanical ventilation or all-cause death
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Anticoagulation | Standard Care
Number analyzed (Participants) | 228 | 237
Participants | 23 | 28

5. Secondary Outcome: Major Bleeding
Description: Major bleeding as defined by the ISTH Scientific and Standardization Committee (ISTH-SSC) recommendation
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Anticoagulation | Standard Care
Number analyzed (Participants) | 228 | 237
Participants | 2 | 4

6. Secondary Outcome: Red Blood Cell Transfusion
Description: Red Blood Cell transfusion (greater than or equal to 1 unit)
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Anticoagulation | Standard Care
Number analyzed (Participants) | 228 | 237
Participants | 3 | 9

7. Secondary Outcome: Transfusion of Platelets, Frozen Plasma, Prothrombin Complex Concentrate, Cryoprecipiate and/or Fibrinogen Concentrate
Description: Transfusion of platelets, frozen plasma, prothrombin complex concentrate, cryoprecipiate and/or fibrinogen concentrate
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Anticoagulation | Standard Care
Number analyzed (Participants) | 228 | 237
Participants | 1 | 0

8. Secondary Outcome: Renal Replacement Therapy
Description: Renal replacement therapy defined as continuous renal replacement therapy or intermittent hemodialysis
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Anticoagulation | Standard Care
Number analyzed (Participants) | 228 | 237
Participants | 2 | 5

9. Secondary Outcome: Hospital-free Days Alive up to Day 28
Description: Hospital-free days alive up to day 28
Time Frame: Up to 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Therapeutic Anticoagulation | Standard Care
Number analyzed (Participants) | 228 | 237
days | 19.8 (7.3) | 18.4 (9.2)

10. Secondary Outcome: ICU-free Days Alive up to Day 28
Description: ICU-free days alive up to day 28
Time Frame: Up to 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Therapeutic Anticoagulation | Standard Care
Number analyzed (Participants) | 228 | 237
days | 26 (6.1) | 24.2 (8.8)

11. Secondary Outcome: Ventilator-free Days Alive up to Day 28
Description: Ventilator-free days alive up to day 28
Time Frame: Up to 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Therapeutic Anticoagulation | Standard Care
Number analyzed (Participants) | 228 | 237
days | 26.5 (5.6) | 24.7 (8.5)

12. Secondary Outcome: Organ Support-free Days Alive up to Day 28
Description: Organ support-free days alive up to day 28
Time Frame: Up to 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Therapeutic Anticoagulation | Standard Care
Number analyzed (Participants) | 228 | 237
days | 25.8 (6.2) | 24.1 (8.8)

13. Secondary Outcome: Venous Thromboembolism
Description: Venous thromboembolism
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Anticoagulation | Standard Care
Number analyzed (Participants) | 228 | 237
Participants | 2 | 6

14. Secondary Outcome: Arterial Thromboembolism
Description: Arterial thromboembolism
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Anticoagulation | Standard Care
Number analyzed (Participants) | 228 | 237
Participants | 0 | 1

15. Secondary Outcome: Heparin Induced Thrombocytopenia
Description: Heparin induced thrombocytopenia
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Anticoagulation | Standard Care
Number analyzed (Participants) | 228 | 237
Participants | 0 | 0

16. Secondary Outcome: Changes in D-dimer
Description: Geometric mean ratio defined as ratio of geometric means of D-dimer ratios (D-dimer×ULN) of day 2 ±24 hours post-randomisation, adjusted for baseline geometric means of D-dimer ratios using analysis of covariance.
Time Frame: Up to day 3
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Therapeutic Anticoagulation | Standard Care
Number analyzed (Participants) | 228 | 237
ratio | 1.9 (0.7) | 2.4 (0.9)

ADVERSE EVENTS:
Time Frame: 28 Days
Arm/Group | Therapeutic Anticoagulation | Standard Care
All-Cause Mortality (participants affected / at risk) | 4/228 | 18/237
Serious Adverse Events (participants affected / at risk) | 228/228 | 237/237
Other Adverse Events (participants affected / at risk) | 228/228 | 237/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Therapeutic Anticoagulation (N=228) | Standard Care (N=237)
Hospitalization (General disorders) | 228 | 237 — Hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Therapeutic Anticoagulation (N=228) | Standard Care (N=237)
Laboratory confirmed SARS-CoV-2 infection (Respiratory, thoracic and mediastinal disorders) | 228 | 237

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT04362085/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT04362085/SAP_001.pdf